CLINICAL TRIAL: NCT02886260
Title: Establishing a Descriptive Cohort of Patients Cared for Operation on the Spine
Acronym: KEOPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2011/PK-01
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Quality of Life; Spinal Injuries; Spinal Diseases
MeSH Terms: conditions — Spinal Injuries; Spinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to:

1. describe the monitoring of patients treated for spinal disorders.
2. create a comprehensive database of reliable and readily exploitable quickly to produce a library of cross publications between orthopedic surgery and neurosurgical services. This database will include clinical, functional , radiographic , educational, social and professional data.
3. obtain a cohort of patients in the comprehensive range of spinal pathologies.
4. standardize data collection in this cohort with similar national projects.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be given free and informed consent and signed the consent
* The patient must be affiliated or beneficiary of a health insurance plan
* The patient is available for a 24-month follow-up
* The patient is at least 18 years old
* The patient has a symptomatic spinal pathology requiring surgical or orthopedic treatment

Exclusion Criteria:

* The patient is under judicial protection, guardianship or curatorship
* The patient refuses to sign the consent
* It is not possible to give informed information to the patient
* The patient does not fluently read French.
* the patient is not available for a 24-month follow-ip

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with symptomatic spinal pathology requiring surgical or orthopedic treatment
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2012-08-28 (Actual); Primary Completion 2017-06-26 (Actual); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Quality of life measured by the Oswestry Disability Index score | 24 months after surgical intervention

SECONDARY OUTCOMES:
Quality of life measured by the Oswestry Disability Index score | 6 weeks, 12 weeks, 6 months, 12 months, 36 months, 48 months after surgical intervention

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nimes, Nîmes, France